CLINICAL TRIAL: NCT02977221
Title: Evaluation of the Efficacy of Flapless Corticotomy Accomplished by Piezosurgery in Accelerating Orthodontic Treatment of Crowding in Adults: a Randomized Controlled Trial
Brief Title: Efficacy of Piezosurgey Corticotomy (a Minimally Invasive Surgical Technique) in Accelerating Orthodontic Alignment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-OMFS-01-2016
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Surgical Incision; Malocclusion
Keywords: corticotomy; piezocision; piezosurgery; acceleration of tooth movement; crowded anterior teeth
MeSH Terms: conditions — Surgical Wound; Malocclusion | interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Piezosurgery (Experimental): Piezosurgery will be performed on the anterior lower segment of the dental arch in order to accelerate the correction of mandibular anterior crowding.
  Interventions: Procedure: Piezosurgery
- Ordinary Alignment (No Intervention): Treatment will be provided to the patients without any surgical interventions.

INTERVENTIONS:
Procedure: Piezosurgery — The device tip will be used to to create small vertical incisions into the cortex of the dento-alveolar process of the lower anterior teeth.
  Other Names: Piezocision
  Arms: Piezosurgery

SUMMARY:
Applying flapless piezocision corticotomies on the alveolar bone and separating anterior mandibular teeth using a piezosurgery device (i.e. ultrasonic waves that perform very accurate incisions without any sutures following this procedure) may improve the speed of tooth alignment during orthodontic treatment. This study consists of two groups, patients will be randomly assigned to one of these two groups. The efficacy of this procedure on 18 patients (experimental group) will be evaluated,whereas the second group (control group) will receive a traditional orthodontic therapy. The time required to achieve complete alignment of crowded mandibular anterior teeth (from canine to canine) will be compared between the two groups.

DETAILED DESCRIPTION:
According to the American Association of Orthodontists (AAO), the length of comprehensive orthodontic treatment ranges between 18-30 months, depending on treatment options and individual characteristics. In addition, orthodontic treatment time ranges between 25-35 months for extraction therapies, respectively. Reducing orthodontic treatment time is one of the main goals for orthodontists, due to problems such as root resorption, periodontal disease and caries that are associated with prolonged treatment time.

Many techniques have been introduced to accelerate orthodontic tooth movement; surgical and non-surgical. The surgical approach is the most clinically applied and most tested with known predictions and stable results. Surgical approaches usually vary from total block osteotomies to flapless partial corticotomies .In spite of corticotomy-assisted orthodontic treatment efficiency, the invasiveness of these procedures (i.e. requiring full mucoperiosteal flaps elevation) might have limited their widespread acceptance among orthodontists and patients. Therefore, more conservative flapless corticotomy techniques have recently been proposed. These procedures can be accomplished in a reasonably short periods that might produce less pain and discomfort, so we will gain better patient acceptance. Although various techniques of flapless corticotomy have been reported to be successful in practice, scientific evidence for their effectiveness so far has been limited to case series and a few clinical trials, generally with small groups. This study aims to provide some evidence about the efficacy of piezosurgery in a flapless technique to align crowded lower anterior teeth using a parallel-group randomized controlled trial study design.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients , Male and female, Age range: 15-27 years.
2. Severe crowding ≤ 7 (Little's irregularity index)
3. Permanent occlusion.
4. Exist all the Mandibular teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth<4 mm
   * No radiographic evidence of bone loss .
   * Gingival index≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, NSAIDs, …)
2. Patients have anti indication for oral surgery ( medical - social - psycho)
3. Presence of primary teeth in the mandibular arch
4. Missing permanent mandibular teeth (except third molars).
5. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
6. Patient had previous orthodontic treatment

Ages: 15 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Duration of tooth alignment | This will be measured at the end of treatment by calculating the time required time (in days) to achieve complete alignment of lower anterior teeth from the first day of treatment and up to 120-150 days of observation
  This outcome will be measured in 'days'.
Change in Tooth Alignment at one month | Little Index of Irregularity will be measured at 30 days after the onset of treatment.
  This index is measured on plaster study casts of patients' teeth. The value obtained will be compared to the value obtained at the beginning of treatment.
Change in Tooth Alignment at two months | Little Index of Irregularity will be measured at 60 days after the onset of treatment.
  This index is measured on plaster study casts of patients' teeth. The value obtained will be compared to the value obtained at the beginning of treatment.
Change in Tooth Alignment at last assessment time | Little Index of Irregularity will be measured when a complete alignment is achieved; this is expected between 90 to 120 days after the onset of treatment.
  This index is measured on plaster study casts of patients' teeth. The value obtained will be compared to the value obtained at the beginning of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Gibreal, DDS, Principal Investigator — MSc student, Oral and Maxillofacial Surgery Department, University of Damascus Dental School; Bassel Brad, DDS MSc PhD, Study Director — Associate Professor of Oral and Maxillofacial Surgery, Department of Oral and Maxillofacial Surgery, Univ. of Damascus Dental School; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, Department of Orthodontics, University of Damascus Dental School
Locations (1):
- Departments of Orthodontics and Oral and Maxillofcial Surgery, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sebaoun JD, Surmenian J, Dibart S. [Accelerated orthodontic treatment with piezocision: a mini-invasive alternative to conventional corticotomies]. Orthod Fr. 2011 Dec;82(4):311-9. doi: 10.1051/orthodfr/2011142. Epub 2011 Nov 23. French. PMID 22105680
- [Background] Vercellotti T, Podesta A. Orthodontic microsurgery: a new surgically guided technique for dental movement. Int J Periodontics Restorative Dent. 2007 Aug;27(4):325-31. PMID 17726988
- [Background] Keser EI, Dibart S. Sequential piezocision: a novel approach to accelerated orthodontic treatment. Am J Orthod Dentofacial Orthop. 2013 Dec;144(6):879-89. doi: 10.1016/j.ajodo.2012.12.014. PMID 24286911
- [Derived] Gibreal O, Hajeer MY, Brad B. Efficacy of piezocision-based flapless corticotomy in the orthodontic correction of severely crowded lower anterior teeth: a randomized controlled trial. Eur J Orthod. 2019 Mar 29;41(2):188-195. doi: 10.1093/ejo/cjy042. PMID 29931294